CLINICAL TRIAL: NCT02971904
Title: Analyzer of Human Milk: Applicability in Clinical Practice in Order to Achieve the Best Nutrition for Infants: Observational Study.
Brief Title: Analyzer of Human Milk: Applicability in Clinical Practice in Order to Achieve the Best Nutrition for Infants
Acronym: MISTU
Status: Completed | Type: Observational
Sponsor: Danone Early Life Nutrition Brazil (Industry)
Collaborators: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: DanoneELN-02
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Low-Birth-Weight Infant; Premature Infants
Keywords: newborn; prematurity; preterm; human milk; human milk analyzer; neonatology; neonatal intensive care unit; low birth weight
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Human milk collection: Lactating mothers should have enough milk to provide enough maternal milk their preterm infant(s) require plus additional collection of samples (3mL). After consenting to the study, milk from lactating mothers of preterm infants in the local ICU will be analyzed daily from the moment they express sufficient milk volume beyond their child's requirement until discharge (from 4th day of admission until 15th day of hospitalization ). Three mL of sample milk will be collected every morning and analyzed, according to hospital routine. Personal details of mothers and their infants will be collected by applying a questionnaire on the first day of analysis. The nutritional composition of the last meal before the milk sample collection and also a nutrition questionnaire intake will be evaluated.
  Interventions: Other: human milk collection

INTERVENTIONS:
Other: human milk collection

SUMMARY:
An observational and prospective study involving about 30 healthy lactating mothers whose preterm infant(s) is/are hospitalized at Neonatal Intensive Care Unit after childbirth and who can provide enough maternal milk (3mL) to be analyzed from 4th day of admission until 15th day of hospitalization or until discharge.

Considering the lack of evidence related to breast milk nutritional composition from Brazilian lactating mothers of preterm infants; and also the utilization of human milk analyzer as a tool to optimize nutritional therapy and reach proper growth and development of preterm babies, this study aim to evaluate the nutritional composition of human milk from lactating mothers of preterm infant during the hospitalization, the infant grow and also the applicability of mid infrared (MIR) human milk analyzer (HMA) as a methodology.

DETAILED DESCRIPTION:
This is an observational and prospective study involving approximately 30 healthy lactating mothers whose preterm infant(s) is/are hospitalized at Neonatal Intensive Care Unit from the Hospital Santa Casa de Misericordia after childbirth. Lactating mothers should have enough milk to provide enough maternal milk their infant(s) require plus additional collection of samples (3mL). After consenting to the study, milk from lactating mothers of preterm infants in the local ICU will be analyzed daily from the moment they express sufficient milk volume beyond their child's requirement until discharge (from 4th day of admission until 15th day of hospitalization ). Three mL of sample milk will be collected every morning and analyzed, according to hospital routine. Characteristics of subjects and details of their premature children, such as gestational age, birth weight (BMI) and birth details (causes of preterm birth, delivery, complications, etc) will be collected by applying a questionnaire on the first day of analysis. The nutritional composition of the last meal before the milk sample collection and also a three no consecutive nutrition questionnaire daily intake will be evaluated.

The determination of the macronutrient content will be made from the use of Human Milk Analyzer MIRIS (MIRIS HMA), Uppsala, Switzerland, properly calibrated. The analyzer is based on the adopted infrared (IR) technology in combination with a patented technology. Sample collection, storage and analysis, as well as equipment conservation, will be carefully followed according to MIRIS protocol. Information about effectiveness, feasibility and equipment costs will also be evaluated. The data obtained by the HMA will be compared to the nutritional composition of human milk and nutritional needs of preterm found in the literature and included in the main guidelines

ELIGIBILITY:
Inclusion Criteria:

* Healthy mothers with hospitalized preterm newborns
* Enough milk to breastfeed their child and donate 3 ml / day for the study
* Being the first sample of milk collected from the 4th day of hospitalization.

Exclusion Criteria:

* Mothers who are not breastfeeding
* Do not have enough milk for collection.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy, stable mothers, mothers of premature infants who were hospitalized at the neonatal ICU of the Santa Casa de Misericórdia after the birth. Mothers should have enough milk to breastfeed their children, and samples will be collected from April to July 2016.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
evolution of the nutritional composition of maternal milk of mothers of premature infants | up to six months
  Maternal milk energy and protein daily analysis by MIRIS (Mid infrared Human Milk Analyzer)

SECONDARY OUTCOMES:
Impact of mother´s diet in the milk composition | up to six months
  Maternal diet questionnaire in admission and daily last meal record before every human milk collection

IPD SHARING:
Plan to Share IPD: Undecided